CLINICAL TRIAL: NCT05563454
Title: A Randomized, Placebo-controlled, Single-blind, Dose Escalation Study to Investigate the Safety, Tolerability, and Pharmacokinetics of BAY 2395840 After Single and Multiple Dose in Japanese Healthy Male Participants
Brief Title: A Study to Learn How Safe the Study Treatment BAY2395840 is, How it Affects the Body and How it Moves Into, Through, and Out of the Body if Given in Single and in Repetitive Doses to Japanese Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 21822
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Diabetic Neuropathic Pain; Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose step 1 (Experimental): Each participant will receive an single dose (SD) of dose 1 of BAY2395840 or matching placebo.
  Interventions: Drug: BAY2395840
- Dose step 2 (Experimental): Each participant will receive an single dose (SD) of dose 2 of BAY2395840 or matching placebo.
  Interventions: Drug: BAY2395840
- Dose step 3 (Experimental): Each participant will receive an single dose (SD) of dose 3 of BAY2395840 or matching placebo.
  Interventions: Drug: BAY2395840
- Dose step 4 (Experimental): Each participant will receive multiple doses (MDs) of dose 3 of BAY2395840 or matching placebo.
  Interventions: Drug: BAY2395840

INTERVENTIONS:
Drug: BAY2395840 — Administration of dosage form 1 under diet 1 condition

SUMMARY:
Researchers are looking for a better way to treat people who have diabetic neuropathic pain (DNP).

DNP is pain due to damage to the nerves in the extremities that can occur in patients with diabetes as a result of blood sugar levels being too high for too long.

BAY2395840 works by blocking specific receptors. A receptor is a protein inside or on the surface of a cell that binds to a specific substance and causes a specific effect in the cell. BAY2395840 specifically blocks so-called bradykinin B1 receptor, whose activation is involved in inflammatory responses. This blockage may help to relieve pain and inflammation.

BAY2395840 has already been studied in clinical studies with European people. However, data for Japanese people are still missing. The participants of this study do not benefit from this study. However, the study will provide information on how to use BAY2395840 in later studies with Japanese people.

The main purpose of this study is to learn how safe the study drug BAY2395840 is and how it affects the body if given in single and in repetitive doses to Japanese healthy male participants.

To answer this question, the researchers will collect and analyze the medical problems the participants have after taking BAY2395840 and that may or may not be related to the study treatments. These medical problems are also known as "adverse events".

In addition, the study team will learn how BAY2395840 moves into, through and out of the body if given in single and in repetitive doses to Japanese healthy male participants. For this, the researchers will collect data on:

* the (average) highest level of BAY2395840 in the blood (also referred to as Cmax)
* the (average) total level of BAY2395840 in the blood (also referred to as AUC) during the treatment period with the study drug on day 1 and for the repetitive dose group only (see below), on day 7.

Subsequently, the study team will compare the data between those participants who received the study drug BAY2395840 (from different dosing groups) and those participants who received placebo. A placebo is a treatment that looks like a medicine but does not have any medicine in it.

All study participants will be randomly (by chance) assigned to 1 of 5 treatment groups. Dependent on the treatment group, the participants will either take:

* a single dose of the lowest, middle and highest BAY2395840 dose (treatment groups 1 to 3)
* repetitive doses of the highest BAY2395840 dose (treatment group 4) or
* placebo (treatment group 5).

The participants will take their treatments as dosage form 1 after diet 1. The treatment period with repetitive doses of BAY2395840 will be 7 subsequent days.

The participants from treatment groups 1 to 3 will have an in house-period of 8 days including 7 overnight stays. The participants from treatment group 4 will have an in house-period of 12 days including 11 overnight stays. The study duration will be approximately 6 weeks per participant for dose groups 1 to 3 and approximately 7 weeks per participant for dose group 4.

During the study, the study team will:

* take blood and urine samples
* do physical examinations
* check the vital signs such as blood pressure, heart rate, body temperature
* examine heart health using electrocardiogram (ECG).

About 10 to 14 days after the participants take their last treatment, the study doctors and their team will check the participants' health.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, vital signs (BP and pulse rate), 12-lead ECG, and laboratory tests. Re-screening will be allowed.
* Ethnicity: Japanese
* Participant must be 20 to 45 years of age inclusive, at the time of signing the informed consent.
* BMI above or equal 18.0 kg/m^2 and below or equal 29.9 kg/m^2 at screening
* Male
* Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Study participants of reproductive potential must agree to use adequate contraception when sexually active. This applies for the time period between signing of the ICF and 90 days after administration of the study intervention. Acceptable methods of contraception include, but are not limited to: (i) condoms (male or female); (ii) intra-uterine device; (iii) hormone-based contraception. Study participants of reproductive potential must agree to utilize 2 reliable and acceptable methods of contraception simultaneously including condoms.
* A sexually active man who has not been surgically sterilized has to agree not to act as sperm donor for the time period between signing of the ICF and 90 days after the last administration of study intervention.

Exclusion Criteria:

* Any findings from the medical examination (including medical history, physical examination, vital signs, laboratory tests, and 12-lead ECG) deviating from normal and deemed to be of clinical relevance by the investigator.
* Relevant diseases within the last 4 weeks prior to first administration of study intervention.
* Known severe allergies.
* Regular use of therapeutic or recreational drugs.
* Suspicion of drug or alcohol abuse.
* Positive cotinine test.
* Donation of more than 200 mL of blood within 4 weeks before first administration of study intervention, donation of more than 400 mL of blood within 3 months before first administration of study intervention, or plasmapheresis within 3 months prior to first administration of study intervention.
* Intake of foods or beverages containing grapefruit, pomelo, tangelo, or Seville oranges from 7 days before first administration of the study intervention up to the last time point of PK sampling after the last administration of the study intervention.
* Special diets preventing the participants from eating the standard meals during the study conduct.
* Participation in a clinical study of an investigational drug within 4 months or of an approved drug within 3 months before the first administration of study intervention.
* Criteria which in the opinion of the investigator preclude participation for scientific reasons, for reasons of compliance, or for reasons of the participant's safety.
* Participant is in custody by order of an authority or a court of law.
* Participant is an employee of the sponsor or of a CRO conducting the study, or has a close affiliation with the investigational site.
* Unable/unwilling to comply with study restrictions.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) | 10 to 14 days after last administration of study intervention

SECONDARY OUTCOMES:
Cmax (maximum observed drug concentration in measured matrix after single dose administration) of BAY2395840 | On day 1
AUC (area under the concentration vs. time curve from zero to infinity after single (first) dose) of BAY2395840 | On day 1
  AUC(0-tlast) will be used if AUC cannot be determined reliably in all participants.
  AUC(0-tlast): AUC from time 0 to the last data point >LLOQ (lower limit of quantification).
AUC(0-24) (AUC from time 0 to 24 h after single dosing) of BAY2395840 | On day 1
Cmax,md (Cmax after MD administration during a dosage interval, directly taken from analytical data) of BAY2395840 (only for Dose step 4) | On day 7
AUC(0-24)md (AUC from time 0 to 24 h after multiple dosing) of BAY2395840 (only for Dose step 4) | On day 7

CONTACTS AND LOCATIONS:
Locations (1):
- SOUSEIKAI Fukuoka Mirai Hospital, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.